CLINICAL TRIAL: NCT06686303
Title: Combined Effects of Segmental Vibrator With Neuromuscular Electrical Stimulation for Flexor and Extensor Muscle Groups on Upper Limb Function in Sub Acute Stroke
Brief Title: Effects of Combined Segmental Vibrator and Neuromuscular Electrical Stimulation in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0216 RabiaSaleem
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Subacute Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received the high frequency segmental vibrator.
  Interventions: Other: High frequency Segmental Vibrator
- Group B (Experimental): Group B received the combined effects of high frequency segmental vibrator and neuromuscular electrical stimulation.
  Interventions: Other: Combined effects of high frequency segmental vibrator and neuromuscular electrical stimulation.

INTERVENTIONS:
Other: High frequency Segmental Vibrator — Segmental vibrations of high frequency was used on each flexor and extensor interspersed with a 1 minute break.
  Arms: Group A
Other: Combined effects of high frequency segmental vibrator and neuromuscular electrical stimulation. — Segmental vibrations of high frequency with Neuromuscular Electrical Stimulation was given on each flexor and extensor.
  Arms: Group B

SUMMARY:
Stroke is leading cause of death and disability worldwide, resulting in significant functional limitations and disabilities experienced by stroke survivors, particularly in the upper limb. There is a need for more effective interventions targeting upper limb sensory motor impairments. The aim of this study is to study combined effect of segmental vibrator and neuromuscular electrical stimulation for flexor and extensor muscle groups on upper limb function in sub-acute stroke.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted in physiotherapy department of Allama Iqbal Memorial Teaching Hospital Sialkot, National Bone and Joint Hospital and Bashir Hospital Sialkot. Forty stroke patients will be recruited through non-probability convenience sampling technique and will be randomly divided in two equal groups Group A and group B through lottery method. Group A will receive high frequency segmental vibration on flexor and extensor muscle groups while group B will receive neuromuscular electrical stimulation along with high frequency segmental vibration(100Hz) on flexor and extensor muscle groups Data will be collected from patients of sub-acute stroke by using screening tool MoCA(for cognition) and assessment tools Fugl-Meyer Assessment Scale(for upper limb function), Wolf Motor Functional Test(for motor function), Modified Ashworth Scale(for spasticity) , Barthel Index(for ADLs), Maximal Hand Grip Strength(for manual dexterity), Maximal Pinch Grip(for manual dexterity), Nottingham Sensory Assessment(for somatosensory function). An informed consent will be taken. Outcome measures will be assessed at baseline, at 4th week and at 8th week. Follow up will be performed at 12th week. Data analysis will be done by SPSS version 28.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Aged between 45 and 65 years old
* First ever ischemic stroke experienced more than 3 months before the enrollment
* Spasticity of spastic agonist muscles ranging from 0-2 on the MAS

Exclusion Criteria:

* Patients with bilateral brain lesions
* Ischemic involvement of cerebellum or basal ganglia
* Psychiatric disease and cognitive impairment
* Previous history of other neurological diseases,rheumatic and orthopaedic conditions
* Patients under anti-spastic therapy or other clinical trials
* Metal implants e.g. cardiac pacemakers

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
MoCA(Montreal Cognitive Assessment) | Baseline and 8 weeks
  MoCA is a screening tool used to evaluate the cognition in stroke patients. Maximum Score 30 Score > 25 considered normal cognition
Fugl-Meyer Assessment | Baseline and 8 weeks
  Fugl-Meyer is an assessment tool used to evaluate the upper limb function in stroke patients. Upper Extrimity Maximum Score: 66
Wolf Motor Functional Test | Baseline and 8 weeks
  Wolf Motor Functional Test is an assessment tool used to evaluate motor function in stroke patients. The WMFT consists of 15 functional tasks and 2 strength-based tasks (total 17 items). Each task is rated on a 6-point ordinal scale
Barthel Index | Baseline and 8 weeks
  BI is an assessment tool used to evaluate ADLs in stroke patients. Minimum Score: 0 (completely dependent) and Maximum Score: 100 (fully independent)
Modified Ashworth Scale | Baseline and 8 weeks
  MAS is an assessment tool used to evaluate spasticity in stroke patients. Minimum score 0 and maximum score 4
Maximal Hand and Pinch Grip Strength | Baseline and 8 weeks
  Maximal Hand and Pinch Grip Strength is an assessment tool used to evaluate manual dexterity in stroke patients measured by Dynamometer.
Nottingham Sensory Assessment | Baseline and 8 weeks
  Nottingham Sensory Assessment is an assessment tool used to evaluate somatosensory sensation in stroke patients. Minimum Score: 0, Maximum Score: 42 (normal sensation)

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- National Bone and Joint Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No